CLINICAL TRIAL: NCT00563433
Title: MSI-78 Topical Cream vs. Oral Ofloxacin in the Treatment of Infected Diabetic Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abeona Therapeutics, Inc (Industry)
Collaborators: Genaera Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI-78-304
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic; diabetes mellitus; foot; ulcers; Floxin; oral antibiotic; topical cream
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Ulcer | interventions — Ofloxacin; pexiganan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ofloxacin (Active Comparator): an oral antibiotic (ofloxacin 400 mg) twice a day and a placebo vehicle topical cream twice a day for 14 days, extended up to 28 days if clinically warranted
  Interventions: Drug: ofloxacin
- MSI-78 (Active Comparator): an oral placebo twice a day and MSI-78 1%/2% Topical Cream twice a day for 14 days, extended up to 28 days if clinically warranted.
  Interventions: Drug: MSI-78

INTERVENTIONS:
Drug: ofloxacin — 400 mg twice a day for 14 days
  Other Names: Floxin
  Arms: ofloxacin
Drug: MSI-78 — 1%/2% topical cream twice a day for 14 days
  Arms: MSI-78

SUMMARY:
224 adults with diabetic foot ulcers will be randomized to either magainin peptide (MSI-78) or ofloxacin (FLOXIN, Ortho-McNeil Pharmaceutical Corporation) an oral fluoroquinolone antibiotic.

DETAILED DESCRIPTION:
Approximately 224 adults will be enrolled in an outpatient Phase III study to compare the safety and efficacy of topically applied magainin peptide (MSI-78) to that of ofloxacin (FLOXIN, Ortho-McNeil Pharmaceutical Corporation) an oral fluoroquinolone antibiotic, in the treatment of infected diabetic foot ulcers.

This is a randomized, controlled, double-blind trial that will involve twenty or more clinical centers.

ELIGIBILITY:
Inclusion Criteria:

* Non-hospitalized ambulatory patients with diabetes mellitus
* Men or Women greater than 18 years old
* Patients must be considered reliable, willing and able to give consent
* Female patients must be postmenopausal for a least 6 months or surgically sterilized
* Localized infection of the ulcer that would ordinarily be treated on an outpatient basis
* Patients who have been previously treated or are currently under treatment for a localized infections of an ulcer may be enrolled in there has been an adequate response to treatment and ulcer is still infected
* Patient must have radiograph within two weeks of entry showing no evidence of cortical destruction consistent with osteomyelitis
* Patient must have a palpable dorsalis pedis or posterior tibial pulse in the affected foot
* Patient may not be taking or have received any other investigational therapy or approved therapy within 30 days prior to entry

Exclusion Criteria:

* Patients requiring concurrent local or systemic antimicrobials during the study period for other infections
* Patients who are currently treated or awaiting dialysis
* Patients who are unable to care for their ulcers
* Patients with known alcohol or substance abuse within 6 months or study entry
* Patients with significant GI problems or surgery that might interfere with the absorption of ofloxacin
* Patients who are currently receiving systemic corticosteroids, immunosuppressives, antivirals, radiation therapy or cytotoxic agents
* Patients who currently require treatment or a primary or metastatic malignancy or have systemically immunocompromising disease.
* Previous enrollment in this study or previous treatment with MSI-78 Topical Cream
* Patients with gangrene or severely impaired arterial supply to any portion of the affected foot
* Other conditions considered by the investigator to be sound reason for disqualification
* Patients with any known allergy to ofloxacin, other quinolone antibiotics, magainin peptides or ingredients of the vehicle cream
* Women who are breast feeding, pregnant or attempting to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 1994-08 (Actual); Primary Completion 1996-07 (Actual); Study Completion 1996-07 (Actual)

PRIMARY OUTCOMES:
Reduction in clinical signs and symptoms of infection | Study day 10
  Measure will be a comparison of the reduction in clinical signs and symptoms of infection between MSI-78 topical therapy and conventional oral antibiotic therapy

SECONDARY OUTCOMES:
Microbiological response | Study day 10
  Measure microbiological response to therapy
Wound infection score | Study day 10
  Measure wound infection score
Total wound score | Study day 10
  Measure total wound score
Wound area | Study day 10
  Measure wound area.
Wound depth. | Study day 10
  Measure wound depth.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Litka, MD, Study Director — Magainin Pharmaceuticals, Inc.
Locations (1):
- Seattle VA Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Lipsky BA, Holroyd KJ, Zasloff M. Topical versus systemic antimicrobial therapy for treating mildly infected diabetic foot ulcers: a randomized, controlled, double-blinded, multicenter trial of pexiganan cream. Clin Infect Dis. 2008 Dec 15;47(12):1537-45. doi: 10.1086/593185. PMID 18990064